CLINICAL TRIAL: NCT00134589
Title: Increasing CRC Screening in Health Plan Members
Brief Title: CHOICE: Communicating Health Options Through Information and Cancer Education
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of North Carolina (Other); Aetna, Inc. (Industry)
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: CDC-NCCDPHP-R-01-PH-000018
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2007-07

CONDITIONS: Colorectal Neoplasms
Keywords: Academic Detailing; Decision Aid; Colorectal Cancer Screening; RECTAL NEOPLASMS; COLONIC POLYPS
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Colonic Polyps

INTERVENTIONS:
Behavioral: Academic Detailing (Medical Practices)+Decision Aids (Patients)

SUMMARY:
The purpose of this study is to determine the effectiveness of a two-component intervention, that combines academic detailing at the medical practice level and distribution of decision aids at the patient level, on adherence to colorectal cancer screening guidelines.

DETAILED DESCRIPTION:
Colorectal cancer is the second most common cause of cancer death in the United States. Early detection and intervention can significantly reduce morbidity and mortality from colorectal cancer (CRC), and current guidelines recommend that asymptomatic adults over age 50 periodically obtain screening by one of several modalities (FOBT, sigmoidoscopy, colonoscopy, or double contrast barium enema). However, CRC screening remains substantially underutilized in the U.S., and more than half of all adults do not adhere to these recommendations. This study was designed to increase CRC screening among health plan members, and involves the collaboration of a major health insurer.

We are conducting a cluster-randomized trial in health practices in Georgia and Florida, to test the effectiveness of a decision aid (video + brochures) for increasing adherence to CRC screening guidelines. Thirty-two large group practices were recruited and randomized to receive usual care (routine reminders) or an evidence-based decision aid intervention. In each practice, patients between the ages of 52 and 75, without current CRC screening history, were enrolled into the study.

In early 2007, we received a full HIPAA waiver that permitted us to send the decision aid intervention to long-term non-responders in the intervention group, and to access claims data for this group and the long-term non-responders in the usual care group. This procedure will make it possible for us to learn more about the real-world impact of the intervention.

The intervention will continue for up to 2 years for still-unscreened participants. The main outcome is receipt of an evidence-based modality of CRC screening according to the US Preventive Services Task Force Guidelines (FOBT, flexible sigmoidoscopy, colonoscopy, or double contrast barium enema).

Unique features of the proposed study include its potential to establish systems to increase screening uptake that will help fulfill HEDIS requirements; improving our understanding of how screening promotion interventions work in both White and Black populations; collaboration with a community partner of the Emory Prevention Research Center, and forging collaborative relationships between public health and health care researchers, and the affected communities of health plans and health care providers.

ELIGIBILITY:
Inclusion Criteria:

* Ages 52-75
* Aetna Health Plan member
* Average risk for colorectal cancer
* Did not have colorectal cancer screening within guideline time frame (1 to 10 years, depending on individual's age and type of screening)

Exclusion Criteria:

* History of colorectal cancer, polyps, inflammatory bowel disease, upper or lower gastrointestinal bleeding, cirrhosis, chronic obstructive pulmonary disease, cancer, blindness, uncorrectable hearing loss, severe dementia, severe heart failure, severe coronary artery disease
* Family history of colorectal cancer/polyps

Ages: 52 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2005-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Completion of colorectal cancer screening

SECONDARY OUTCOMES:
Patient's intention to ask/patient asking medical provider for colorectal cancer screening

CONTACTS AND LOCATIONS:
Overall Officials: Karen Glanz, PhD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory University Rollins School of Public Health, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Pignone M, Winquist A, Schild LA, Lewis C, Scott T, Hawley J, Rimer BK, Glanz K. Effectiveness of a patient and practice-level colorectal cancer screening intervention in health plan members: the CHOICE trial. Cancer. 2011 Aug 1;117(15):3352-62. doi: 10.1002/cncr.25924. Epub 2011 Feb 11. PMID 21319147
- [Derived] Pignone M, Scott TL, Schild LA, Lewis C, Vazquez R, Glanz K. Yield of claims data and surveys for determining colon cancer screening among health plan members. Cancer Epidemiol Biomarkers Prev. 2009 Mar;18(3):726-31. doi: 10.1158/1055-9965.EPI-08-0751. PMID 19273480